CLINICAL TRIAL: NCT00197392
Title: Establishment of Baseline and Comparative Infection Rates for the Codman BACTISEAL TM External Ventricular Drainage (EVD) System
Brief Title: Comparative Infection Rates for the Codman BACTISEAL TM External Ventricular Drainage (EVD) System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAC-IN02-002
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Intraventricular Hemorrhage; Subarachnoid Hemorrhage
Keywords: Ventriculostomy; EVD
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bactiseal TM EVD (Experimental): Bactiseal External Ventricular Drainage System.
  Interventions: Device: Bactiseal TM EVD
- Standard EVD Catheter (Active Comparator): Standard External Ventricular Device system
  Interventions: Device: Standard EVD Catheter

INTERVENTIONS:
Device: Bactiseal TM EVD — Standard of care implantation of external ventricular drainage catheter
  Other Names: EVD,Bactiseal, standard
  Arms: Bactiseal TM EVD
Device: Standard EVD Catheter — Standard of care EVD system other than Bactiseal.
  Other Names: EVD, ventricular catheters
  Arms: Standard EVD Catheter

SUMMARY:
The purpose of this non-significant risk study is to establish initial baseline infection rates for the Codman BACTISEAL External Ventricular Drainage (B-EVD) System (Antibiotic impregnated catheter) and to compare relative rates of ventriculostomy-related infection between Subjects with BACTISEAL or conventional EVD catheters in a prospective, randomized open label study

DETAILED DESCRIPTION:
External ventricular drainage catheters are widely used in the management of Subjects with elevated intra-cranial pressure (ICP) secondary to acute hydrocephalus due to sub-arachnoid hemorrhage, intra-cerebral hemorrhage, intra-ventricular hemorrhage and other causes that obstruct the cerebrospinal fluid (CSF) circulation. However, this mode of treatment could be compromised by the increased risk of catheter related CSF infection.

B-EVD is manufactured using a patented process to impregnate silicone catheters with two antibiotics, rifampin and clindamycin. These antibiotics are impregnated throughout the silicone matrix. After implantation, slow release of both antibiotics at the extra- and intra-luminal catheter surfaces minimizes the likelihood of bacterial colonization. The B-EVD Catheter System has, to date, been well accepted by domestic and European customers. Currently there exists sound scientific rationale and promising bench-top in vitro data to anticipate low levels of ventriculostomy-related infection in Subjects using this system. Published BACTISEAL shunt data and direct feedback from U.S. market experience also support this notion. There are no published clinical studies reporting infection rates with the use of the B-EVD System, making all statements regarding its propensity to minimize clinical risk for catheter-related infection mere speculation and anecdotal. Therefore, Codman proposes to undertake a controlled clinical evaluation of this product to demonstrate its influence on EVD catheter-related infections, using a conventional EVD catheter as a standard of reference.

Immediately following successful screening, the Subject will be randomized to test or control group and will have the appropriate EVD system implanted. The Treatment Phase will cover the duration of the implanted EVD system. Subjects will be monitored for 2 weeks post-explant.

This study is expected to enroll 600 evaluable implanted Subjects at up to 15 Investigational Sites in US, Europe and Asia-Pacific

ELIGIBILITY:
Inclusion Criteria:

* The Subject is 18 years or older.
* The Subject (family member/legal representative) has given written Informed Consent prior to enrollment into this trial OR, where the Subject is unable to consent and no relative/legal representative is available to offer consent, appropriate legal and ethical practices are employed and thoroughly documented according to the laws and policies of the respective country and institution.
* The Subject (family member/legal representative) is willing to participate in this trial for the duration of the implanted EVD system and is willing to comply with the protocol requirements.

Exclusion Criteria:

* Within the preceding 30 days, the Subject has enrolled or participated in another trial utilizing an anti-microbial drug or medical device implanted in or directly influencing the CNS and/or spinal cord.
* The Subject is pregnant or lactating.
* The Subject has a suspected or documented allergy to the materials of the EVD system, including silicone, rifampin and clindamycin.
* The Subject has a positive CSF culture prior to EVD implant.
* The Subject is immunocompromised.
* The Subject requires more than one ventricular catheter concurrently.
* The Subject has had an EVD catheter within the previous 30 days.
* The Subject has sepsis, ventriculitis, meningitis, a skin infection/inflammation at or near the implantation site, an ear infection on either side, or a severe respiratory tract infection that, in the opinion of the Investigator, would most likely compromise the effectiveness of the EVD system.
* The Subject is known to have received systemic antibiotic therapy within a 14-day period preceding screening for inclusion in this trial.
* The Subject has an uncontrolled coagulopathy or any other known bleeding diathesis.
* The Subject is otherwise determined by the Investigator to be medically unsuitable for participation in this trial.
* The Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Thomas Megerian, MD, PhD, Study Director — Unaffilliated
Locations (20):
- United States (4):
  - Los Angeles, California
  - Gainesville, Florida
  - Syracuse, New York
  - Hershey, Pennsylvania
- Canada (3):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Sherbrooke, Quebec
- China (2):
  - Tiantan Hospital, Beijing
  - Xuan Wu Hospital, Beijing
- France (3):
  - Angers
  - Lille
  - Paris
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Oslo, Norway
- Singapore (2):
  - National Neuroscience Institute, Singapore
  - Singapore General Hospital, Singapore
- United Kingdom (3):
  - Bristol
  - Leeds
  - Salford

REFERENCES:
- [Background] Codman in house testing reports, TR2213 and PVER99-133 Addendum
- [Background] Bayston R. Hydrocephalus Shunt Infections. Chapman and Hall Medical, London, 1989, p. 23.
- [Background] Bayston R, Grove N, Siegel J, Lawellin D, Barsham S. Prevention of hydrocephalus shunt catheter colonisation in vitro by impregnation with antimicrobials. J Neurol Neurosurg Psychiatry. 1989 May;52(5):605-9. doi: 10.1136/jnnp.52.5.605. PMID 2732730
- [Background] Bayston R, Lambert E. Duration of protective activity of cerebrospinal fluid shunt catheters impregnated with antimicrobial agents to prevent bacterial catheter-related infection. J Neurosurg. 1997 Aug;87(2):247-51. doi: 10.3171/jns.1997.87.2.0247. PMID 9254088
- [Background] Govender ST, Nathoo N, van Dellen JR. Evaluation of an antibiotic-impregnated shunt system for the treatment of hydrocephalus. J Neurosurg. 2003 Nov;99(5):831-9. doi: 10.3171/jns.2003.99.5.0831. PMID 14609161
- [Background] Lozier AP, Sciacca RR, Romagnoli MF, Connolly ES Jr. Ventriculostomy-related infections: a critical review of the literature. Neurosurgery. 2002 Jul;51(1):170-81; discussion 181-2. doi: 10.1097/00006123-200207000-00024. PMID 12182415
- [Background] Schierholz J, Jansen B, Jaenicke L, Pulverer G. In-vitro efficacy of an antibiotic releasing silicone ventricle catheter to prevent shunt infection. Biomaterials. 1994 Oct;15(12):996-1000. doi: 10.1016/0142-9612(94)90080-9. PMID 7841297
- [Background] Zabramski JM, Whiting D, Darouiche RO, Horner TG, Olson J, Robertson C, Hamilton AJ. Efficacy of antimicrobial-impregnated external ventricular drain catheters: a prospective, randomized, controlled trial. J Neurosurg. 2003 Apr;98(4):725-30. doi: 10.3171/jns.2003.98.4.0725. PMID 12691395

RESULTS

PARTICIPANT FLOW:
Groups:
- Bactiseal EVD: Subjects treated with Bactiseal EVD catheter
- Conventional EVD Catheter: Subjects treated with Standard EVD catheter
Period: Overall Study
Arm/Group | Bactiseal EVD | Conventional EVD Catheter
Started | 214 | 220
Safety Population | 214 | 220
Modified Intent to Treat | 209 | 210
Evaluable | 176 | 181
Per Protocol | 126 | 134
Completed | 126 | 134
Not Completed | 88 | 86

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bactiseal EVD | Standard EVD | Total
Number analyzed (Participants) | 214 | 220 | 434
Age Continuous [Mean (Standard Deviation); unit: years] | 51.7 (16.2) | 54.4 (14.7) | 53.05 (15.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 110 | 220
  Male | 104 | 110 | 214
Region of Enrollment [Number; unit: participants]
  France | 30 | 29 | 59
  United States | 36 | 42 | 78
  Hong Kong | 27 | 33 | 60
  Canada | 21 | 17 | 38
  Singapore | 14 | 11 | 25
  Norway | 30 | 26 | 56
  China | 18 | 17 | 35
  United Kingdom | 38 | 45 | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Infections
Description: The number of infections for the Codman Bactiseal EVD Catheter and the number of infections for a Standard EVD Catheter (ventriculostomy-related infections).
Time Frame: Duration of implanted EVD system to 2 week post implant
Measure: Number; unit: Infections
Groups:
- Bactiseal EVD Catheter: Patients treated with Codman Bactiseal EVD Catheter
- Standard EVD Cathter: Patients treated with Standard EVD Catheter
Arm/Group | Bactiseal EVD Catheter | Standard EVD Cathter
Number analyzed (Participants) | 209 | 210
Infections
  Modified intent to Treat | 4 | 5
  Evaluable | 4 | 5
  Per Protocol | 1 | 3

2. Secondary Outcome: Days to Proven Infection
Description: Number of days to proven infection.
Time Frame: Implantation of EVD System to explant of EVD catheter, an average of ten days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Standard EVD Catheter: Patients treated with standard EVD catheter.
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 214 | 220
Days
  Modified Intent to Treat | 9.5 (3.3) | 10 (3.0)
  Evaluable | 9.5 (3.3) | 10 (3.0)
  Per protocol | 14 (1) | 10 (2.5)

3. Secondary Outcome: Class of Bacterial Agent Causing Proven Infection
Description: Type of bacterial agent related to proven infection in Bactiseal EVD and Standard EVD
Time Frame: Implantation of subject to post implant
Population: All subjects included in the MITT, Evaluable and Per-Protocol population.
Measure: Number; unit: participants
Groups:
- Bactiseal - EVD Catheter: Patients treated with Bactiseal EVD catheter
- Standard EVD Catheter: Patient treated with Standard EVD Catheter
Arm/Group | Bactiseal - EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 22 | 22
participants
  Bacilli | 11 | 0
  Gamma Proteobacteria | 0 | 6

4. Secondary Outcome: Intraluminal Colonization on Catheters
Description: Number of catheters with Bacterial colonization verified using fluorescence.
Time Frame: Implant of subjects to post implant
Measure: Number; unit: catheters
Groups:
- Bactiseal EVD Catheter: Patients implanted with Bactiseal EVD Catheter
- Standard EVD Catheter: Patients implanted with Standard EVD Catheter
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 209 | 210
catheters | 0 | 3

5. Secondary Outcome: Device Related Adverse Events
Description: Number of Device Related Adverse Events
Time Frame: Implanted subjects to time of explant
Population: There were 8 device-related events, 7 of which were in subjects that received a standard catheter. None of the 8 subjects were proven infections.
Measure: Number; unit: events
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 214 | 220
events
  Modifeid Intent to Treat | 0 | 1
  Evaluable | 1 | 4
  Per protocol | 0 | 0
  Safety | 0 | 2

6. Secondary Outcome: Number of Days With Indwelling Catheter
Description: Days catheter was implanted in subjects
Time Frame: Implant of subjects to day of explant
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 192 | 199
Days
  Modified Intent to Treat | 8.7 (5.7) | 8.9 (6.0)
  Evaluable | 9.3 (5.5) | 9.7 (5.8)
  Per Protocol | 9.8 (5.7) | 10.4 (5.9)

7. Secondary Outcome: Average Subject Age
Description: The average subject age
Time Frame: Implant to subject
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Bactiseal EVD Catheter: Subjects implanted with Bactiseal EVD Catheter
- Standard EVD Catheter: Subjects implanted with standard EVD catheter
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 209 | 210
Years
  Modified Intent to Treat | 51.9 (16.1) | 54.4 (14.7)
  Evaluable | 51.9 (16.1) | 54.5 (14.6)
  Per protocol | 49.4 (15.8) | 54.2 (14.2)

8. Secondary Outcome: Diagnosis Requiring EVD Implantation
Description: Primary diagnosis for implantation of EVD system
Time Frame: Implantation of EVD system
Population: Analysis consisted of combining both Arm/Group (Bactiseal and Standard)
Measure: Number; unit: Participants
Groups:
- Bactiseal EVD Catheter and Standard EVD Cathter: Patients implanted with Bactiseal EVD Catheter or Standard EVD Catheter.
Arm/Group | Bactiseal EVD Catheter and Standard EVD Cathter
Number analyzed (Participants) | 419
Participants
  Edema - Modified Intent to Treat | 20
  Edema - Evaluable | 17
  Edema - Per Protocol | 13
  Hemorrhage - Modified Intent to Treat | 335
  Hemorrhage - Evaluable | 282
  Hemorrhage - Per protocol | 197
  Hydrocephalus - Modified Intent to Treat | 64
  Hydrocephalus - Evaluable | 58
  Hydrocephalus - Per Protocol | 50

9. Secondary Outcome: Non-infectious Catheter Failure in the MITT Population
Description: Reasons for non-infectious catheter malfunctions in the Modified intent to treat population.
Time Frame: Implant of subject to explant
Measure: Number; unit: Participants
Groups:
- Bactiseal EVD Catheter: Subjects treated with Bactiseal EVD Catheter
- Standard EVD Catheter: Subjects treated with standard EVD catheter
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 176 | 181
Participants
  Occlusion | 16 | 0
  Migration | 0 | 1
  Misplacement | 0 | 1
  Other | 0 | 3

10. Secondary Outcome: Time Point of Introduction of Systemic Antibiotic Therapy
Description: Time points of then patients received systemic antibiotic therapy
Time Frame: Within 48 hours of implant of subjects to explant
Measure: Number; unit: Paticipants
Groups:
- Standrad EVD Catheter: Subjects implanted with standard EVD catheter
Arm/Group | Bactiseal EVD Catheter | Standrad EVD Catheter
Number analyzed (Participants) | 209 | 210
Paticipants
  Before implant, but within 48 hours (MITT) | 146 | 149
  Catheter Implanted (MITT) | 167 | 175
  Before implant, but within 48 hours (Evaluable) | 118 | 124
  Catheter Implanted (Evaluable) | 150 | 159
  Before implant, but within 48 hours (Per protocol) | 81 | 90
  Catheter implanted (Per Protocol) | 108 | 121

11. Secondary Outcome: Hospital Locations for EVD Catheter Placement
Description: Number of subjects in each analysis population where the EVD catheter placement occurred; either in the Intensive Care Unit (ICU)or the Operating Room (OR).
Time Frame: Implantation of subject
Measure: Number; unit: Participants
Groups:
- Bactiseal EVD Catheter: Subjects implanted with the Bactiseal EVD Catheter
- Standard EVD Catheter: Subjects implanted with a standard EVD catheter
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 214 | 220
Participants
  ICU (MITT) | 45 | 49
  OR (MITT) | 159 | 153
  ICU (Evaluable) | 37 | 41
  OR (Evaluable) | 136 | 132
  ICU (Per Protocol) | 22 | 25
  OR (Per Protocol) | 103 | 106

12. Secondary Outcome: Length of Catheter Tunneling Into the Brain
Description: Length of tunneling of EVD catheter in the brain for each analysis population.
Time Frame: Implant of subject
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bactiseal EVD Catheter | Standard EVD Catheter
Number analyzed (Participants) | 202 | 205
cm
  MITT | 6.2 (2.2) | 5.8 (2.1)
  Evaluable | 6.2 (2.1) | 5.8 (2.1)
  Per Protocol | 6.0 (1.9) | 5.7 (1.8)

13. Secondary Outcome: Number of Catheter Insertion Attempts
Description: Number of insertions needed to place catheter
Time Frame: Implantation of subject
Measure: Number; unit: insertions
Groups:
- Bactiseal EVD: Subjects implanted with Bactiseal EVD catheters.
- Standard EVD: Subjects implanted with Standard EVD catheters.
Arm/Group | Bactiseal EVD | Standard EVD
Number analyzed (Participants) | 206 | 208
insertions
  1 Insertion | 177 | 178
  2 insertions | 15 | 16
  3 instertions | 9 | 11
  4 instertions | 3 | 2
  5 insertions | 2 | 1

ADVERSE EVENTS:
Groups:
- Standard EVD: Subjects with standard EVD
- Bactiseal EVD: Subjects with Bactiseal EVD
Arm/Group | Standard EVD | Bactiseal EVD
Serious Adverse Events (participants affected / at risk) | 16/220 | 14/214
Other Adverse Events (participants affected / at risk) | 11/220 | 19/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard EVD (N=220) | Bactiseal EVD (N=214)
Death (Surgical and medical procedures) | 1 (1) | 0 (0)
Sepsis secondary to pneumonia with complicating head injury (Infections and infestations) | 0 (0) | 1 (1)
Respiratory culture positive for staphylocccus (Infections and infestations) | 3 (3) | 1 (1)
Respiratory culture positive for enterobateraerogenes (Infections and infestations) | 1 (1) | 2 (2)
Brain Death (Nervous system disorders) | 0 (0) | 2 (2)
Respiratory culture positive for haemophilus influenzae (Infections and infestations) | 0 (0) | 1 (1)
Respiratory culture positive for staphylocccus aureus-oxacillan resistant (orsa) (Infections and infestations) | 0 (0) | 1 (1)
Throat culture positive for enterobacter aerogenes (Infections and infestations) | 1 (1) | 0 (0)
Nares culture positive for oxacillan resistant staphylocccus aureus (Infections and infestations) | 1 (1) | 0 (0)
CSF positive for coccidiodes immitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory culture positive for escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
CSF culture positive for coagulase negative staphylococcus (Infections and infestations) | 1 (1) | 0 (0)
Epidural hematoma at ventriculostomy site (Infections and infestations) | 0 (0) | 1 (1)
CSF infection (Infections and infestations) | 1 (1) | 2 (2)
CSF infection with secondary hydrocephalus (Infections and infestations) | 1 (1) | 0 (0)
Right intracerebral hemorhage (Cardiac disorders) | 1 (1) | 0 (0)
Aseptic Inflammation (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Ventriculitis (Nervous system disorders) | 0 (0) | 1 (1)
Blood Culture Positive for Coagulase Negative Staphylococcus (Infections and infestations) | 2 (2) | 1 (1)
Vasovagal Shock at EVD Explant (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard EVD (N=220) | Bactiseal EVD (N=214)
Blood positive for streptococcus (Infections and infestations) | 0 (0) | 1 (1)
CNS Infection (Infections and infestations) | 2 (2) | 4 (4)
Coagulase negative staphylococcus in CSF (Infections and infestations) | 1 (1) | 1 (1)
Confirmed dipthroid infection in CSF (Infections and infestations) | 1 (1) | 0 (0)
CSF culture positive for coagulase negative staphylococcus (Infections and infestations) | 1 (1) | 0 (0)
CSF Positive for propionibacterium (Infections and infestations) | 1 (1) | 2 (2)
CSF infection - entermococcus faecacil acinetobacter banmanii (Infections and infestations) | 1 (1) | 0 (0)
CSF Infection - pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Catheter tip - cultutre positive for coagulase negative staphylococcus (Infections and infestations) | 1 (1) | 0 (0)
Catheter occlusion due to hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Increrased intra-cranial pressure (Nervous system disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Sputum culture positive with gram positive cocci & gram negative diplococci (Infections and infestations) | 0 (0) | 1 (1)
Sputum positive for gram negative & gram positive rods (Infections and infestations) | 0 (0) | 1 (1)
Sputum positive for staphylococcus (Infections and infestations) | 0 (0) | 1 (1)
Stomach Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Trubid CSF (Surgical and medical procedures) | 0 (0) | 1 (1)
Urine positive for escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Vasovagal Shock (Nervous system disorders) | 1 (1) | 0 (0)
Sputum Positive for Staphylococcus (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days